CLINICAL TRIAL: NCT00280345
Title: Autoimmune Dysregulation in Pigmentary Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pigmentary Glaucoma
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pigmentary Glaucoma; Primary Open Angle Glaucoma; Cataract
Keywords: pigmentary glaucoma; primary open angle glaucoma; cataract; trabeculectomy; cataract surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Trabeculectomy; Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Trabeculectomy — A surgical procedure used in the treatment of glaucoma to relieve intraocular pressure by removing part of the eye's trabecular meshwork
Procedure: Trabeculectomy and cataract surgery — A surgical procedure used in the treatment of glaucoma to relieve intraocular pressure by removing part of the eye's trabecular meshwork and the removal of the cataract
Procedure: Cataract surgery — Removal of the cataract from the eye

SUMMARY:
Based on these recent observations and findings in this new animal model of pigmentary glaucoma in the DBA/2J mouse, we propose that immune system abnormalities in the anterior chamber may play a possible role in the development of pigmentary glaucoma and possibly primary open-angle glaucoma (POAG) in humans.

DETAILED DESCRIPTION:
The aim is to establish, through tissue and aqueous analysis of patients with pigmentary glaucoma, POAG and normal controls, that markers for anterior chamber autoimmune dysfunction occur in significantly different amounts in patients with these conditions when compared to normal controls. We also will attempt to establish, through proven methodologies of tissue gene expression, that the source of these differences in markers, notably PEDF and IL-18, is from the uveal tissues of the anterior chamber, most importantly the iris and possibly the trabecular meshwork as well.

The actual etiology at the cellular level of elevated intraocular pressure and the development of pigmentary glaucoma is not well understood in humans. If anterior chamber immune dysfunction were shown to be an important factor in the development of this disease in humans, which apparently is demonstrated by the DBA/2J mouse, it would lead to an important area of further investigation and possible novel approaches in treating or preventing this disease in humans.

We hypothesize that in patients with pigmentary glaucoma, the amount of PEDF in the aqueous is significantly reduced while IL-18 is significantly elevated when compared to the aqueous of normal controls. In patients with POAG, we hypothesize similar results for PEDF, although significantly less reduction of PEDF when compared to the pigmentary glaucoma patients may be an interesting finding as well. With regard to IL-18, it is possible that amounts would be significantly elevated in the pigmentary glaucoma patients when compared to both normal controls and POAG patients. In view of the results from the DBA/2J mouse model, we hope to determine whether expression of PEDF could be down regulated in the iris and/or trabecular meshwork of pigmentary glaucoma patients when compared to POAG patients and whether IL-18 expression in these tissues could be up regulated in pigmentary glaucoma patients when compared to POAG patients.

Such findings would strongly suggest that anterior chamber immune abnormalities play a role in the etiology of pigmentary glaucoma in humans. It already has been suggested that decreased amounts and expression of PEDF are found in patients with glaucoma and other neurodegenerative diseases of the eye. However, the source of the decreased expression has not been identified. If IL-18 production is elevated in pigmentary glaucoma and is up regulated in the anterior chamber structures of the eye in human patients with the disease, this also would be highly suggestive that localized anterior chamber immune dysfunction plays a role in the development of this disease.

Depending on our findings, additional investigations of autoimmune dysregulation in pigmentary glaucoma (and perhaps other secondary glaucomas) may help determine the predictive value of such markers in identifying whether or not patients with pigment dispersion syndrome develop glaucomatous damage.

ELIGIBILITY:
Patients in the study will be between 18 and 85 years old. To prevent any possibility that previous manipulation of the iris and uveal structures may affect results of the assays, patients with any previous intraocular surgery or laser iridotomies will be excluded. Patients who have undergone laser trabeculoplasty within 90 days of surgery also will be excluded. In the normal controls undergoing cataract surgery, patients with signs of pigment dispersion syndrome or exfoliation syndrome without glaucoma will be excluded from the study.

Additional Inclusion Criteria:

1. In the glaucoma patients, visual field and/or optic disc changes characteristic of glaucoma.
2. Ability to comprehend the information describing the clinical study.
3. Ability to provide signed and dated IRB-approved informed consent (ICF) for the study.

Exclusion Criteria:

1. Any clinically significant uncontrolled medical condition(s) that might, in the investigators' opinion, interfere with the assessment.
2. Use of corticosteroids within 3 months prior to surgery.
3. Use of systemic anti-metabolites within 6 weeks prior to surgery.
4. Use of any investigational drug within 4 weeks prior to surgery.

Specific to the study eye exclusions:

1. History of non-iatrogenic uveitis or active uveitis.
2. Discernible congenital abnormality of the anterior chamber structures.
3. Neovascular, uveitic, traumatic, or infantile glaucoma.
4. Proliferative or severe non-proliferative diabetic retinopathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Autoimmune Dysergulation in Pigmentary Glaucoma | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Crystal McAfee, MA-HHSA, Study Director — Dean A. McGee Eye Institute
Locations (1):
- Dean A. McGee Eye Institute, Oklahoma City, Oklahoma, United States